CLINICAL TRIAL: NCT02516124
Title: Autologous Stem Cell Transplantation for Progressive Systemic Sclerosis: a Prospective Non-Interventional Approach Across Europe (NISSC) for the Autoimmune Diseases Working Party of the EBMT
Brief Title: EBMT ADWP Prospective Non Interventional Study : AutoHSCT in SSc Patients
Acronym: NISSC
Status: Completed | Type: Observational
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Responsible Party: Sponsor
Other Study IDs: NCT02516124; NCT02264405 (obsolete NCT alias)
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2017-07

CONDITIONS: Autoimmune Diseases
Keywords: Autoimmune diseases; Systemic sclerosis; Autologous Hematopoietic stem cell transplant
MeSH Terms: conditions — Autoimmune Diseases; Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NISSC: Autologous HSCT
  Interventions: Procedure: Autologous HSCT

INTERVENTIONS:
Procedure: Autologous HSCT — 1st AHSCT

SUMMARY:
The purpose of this study is to assess the effectiveness of Autologous Hematopoietic Stem Cell transplantation (AHSCT) for early severe or rapidly progressive Systemic Sclerosis (SSc) as currently performed by different study protocols used across Europe in various EBMT centres through the careful recording and analysis of routinely collected clinical and biological data.

DETAILED DESCRIPTION:
Different protocols are used in the different centres, it is not yet clear which approach will be the most efficient and the safest. Every centre will follow its own local protocol for AHSCT which usually refers to the recent update of the EBMT Guidelines for HSCT in autoimmune disease. Patient selection for AHSCT treatment technique with regard to the risk/benefit balance has to be carefully addressed by standard patient pretransplant evaluation, whereas treatment local regimen, follow-ups evaluation, supportive medication and prophylaxis will be recorded and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Autologous HSCT
* Age between 18 and 65 years at time of transplant.
* Established diagnosis of progressive systemic sclerosis according to ARA-criteria

Exclusion Criteria:

* Pregnancy or inadequate contraception
* Severe concomitant disease
* Reduced lung function
* Previously damaged bone marrow
* Uncontrolled severe infection
* Severe concomitant psychiatric illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with autologous HSCT for severe systemic sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2012-12; Primary Completion 2018-01 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 2 year post transplant
  Progression free survival (PFS), defined as survival since Baseline (the 1st day of mobilisation) without evidence of progression of SSc.

SECONDARY OUTCOMES:
Safety assessed by Treatment related toxicity throughout the study period using WHO toxicity parameters (expressed as maximum grade toxicity per organ system, see appendix) | 2 year post transplant
  Incidence of Adverse Events (AE) and Serious Adverse Events (SE) Neutrophil and platelet engraftment, defined as first day after transplantation with absolute neutrophil count > 500 cells/μL and >20.000 platelets/μL without platelet transfusion, respectively
Overall Survival | 2 year post transplant
  Overall Survival
Response to treatment | at 1 year post transplant
  Response to treatment within 1 year following autologous HSCT, defined as
  * 25% improvement in mRSS (modified Rodnan Skin Score) and/or
  * ≥10% improvement in Diffuse Capacity for carbon monoxide (DLCO) or Forced Vital Capacity (FVC) as compared to baseline without need of further immunosuppression
Improvement in Quality of life | 2 year post transplant
  Assessed by SHAQ (Scleroderma Health Assessment Questionnaire) evolution
Relapse incidence | 2 year post transplant
  Defined as any of the following changes after prior response to treatment on quarterly follow up as defined below:
  * Worsening of mRSS > 25%
  * New/Worsening of organ manifestation: lungs, heart or kidney
100-day Treatment related mortality | 100 days post transplant
  any death during 100 day following transplant that cannot be attributed to progression or relapse of the disease

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Farge, PhD, Study Chair — EBMT ADWP
Locations (1):
- Badoglio Manuela- EBMT Paris Office, Paris, France

REFERENCES:
- [Derived] Henes J, Oliveira MC, Labopin M, Badoglio M, Scherer HU, Del Papa N, Daikeler T, Schmalzing M, Schroers R, Martin T, Pugnet G, Simoes B, Michonneau D, Marijt EWA, Lioure B, Olivier Bay J, Snowden JA, Rovira M, Huynh A, Onida F, Kanz L, Marjanovic Z, Farge D. Autologous stem cell transplantation for progressive systemic sclerosis: a prospective non-interventional study from the European Society for Blood and Marrow Transplantation Autoimmune Disease Working Party. Haematologica. 2021 Feb 1;106(2):375-383. doi: 10.3324/haematol.2019.230128. PMID 31949011
- See also: Organisation website — http://ebmt.org